CLINICAL TRIAL: NCT06072989
Title: A Single Arm, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of B4T2-001 CAR-T in Patients With Advanced Solid Tumors
Brief Title: Repeat Intravenous Infusions of B4T2-001 CAR-T Without Lymphodepleting Chemotherapy for Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Bio4T2 LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4T2-PRC IIT-001
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B4T2-001 CAR T (Experimental): Single Arm and Open Label study consisting of dose escalation study design followed by dose expansion phase at determined MTD.
  Interventions: Biological: B4T2-001 autologous CAR-T

INTERVENTIONS:
Biological: B4T2-001 autologous CAR-T — Each subject will receive multiple intravenous infusions of B4T2-001 autologous CAR-T without preparative chemotherapy (lymphodepletion)

SUMMARY:
This is an open-label, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of autologous B4T2-001 CAR-T in subjects with advanced solid tumors including but not limited to advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma, advanced pancreatic cancer, advanced non-small cell lung cancer (NSCLC), colorectal cancers (CRC) and metastatic breast cancer that tests positive for BT-001 target antigen according to Immunohistochemistry (IHC). The trial builds off first-in-human results from pilot study per clinicaltrials.gov ID: NCT05621486 to administer multiple infusions of B4T2-001 CAR-T without the need to give preparative chemotherapy (lymphodepletion).

DETAILED DESCRIPTION:
This is an open-label dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of lentiviral transduced autologous B4T2-001 CAR-T at up to four Dose Levels. Each treatment Block is composed of three Cycles of B4T2-001 CAR-T administered every 21 days by intravenous route without preparative chemotherapy (lymphodepletion). Subjects with advanced solid tumors will be enrolled. One or more Cycle(s) will be delayed as part of routine dosing plan until (i) absolute neutrophil count (ANC) greater than lower limit of normal (LLN) and (ii) resolution of grade >2 toxicity probably or definitely attributed to prior CAR-T and (iii) CAR-T available. Cycles will discontinue if (i) confirmatory imaging shows progressive disease (PD) and/or (ii) CAR-T cells are unavailable. Each additional Block(s) to begin at least 21 days after third Cycle of prior Block. The next patient(s) may be enrolled at least 21 days after completion of first Cycle of prior patient. The decision for dose escalation decision depends on the safety of first Cycle. Two subjects will be enrolled into each Dose Level. If none experiences a dose-limiting toxicity (DLT), the next cohort of two subjects will be enrolled into the next higher dose level. If a DLT is observed in one subject, four additional subjects will be added into the same dose level. If no additional DLT occur, DL will be escalated to the next higher dose level. If DLT occurs in two or more subjects among two to six subjects at a given dose level, dose escalation will be stopped, and the prior dose level will be expanded to six subjects to confirm maximum tolerated dose (MTD). If there is no more than one subject who experiences a DLT among those six subjects, that dose level is considered the MTD. Response to the treatment will be assessed before and after each Block. CT or MRI or PET for response assessment is anticipated every 60 days till day 180, then every 90 days till the end of the study. If complete response (CR), PD, or partial response (PR) on Day 60's assessment, another imaging study will be performed to confirm findings about 4 weeks later. The tumor marker(s) should be performed at the beginning and end of each Cycle All subjects will receive B4T2-001 CAR-T infusion at a healthcare facility, followed by frequently monitoring at a healthcare facility for at least 7 days to monitor for signs and symptoms of cytokine release syndrome (CRS) including immune effector cell-associated neurotoxicity syndrome (ICANS) and/or hemophagocytic lymphohistiocytosis (HLH) and macrophage activation syndrome (MAS). One dose of tocilizumab will be administrated on Day 7 of each Cycle as prophylaxis for CRS. The study follows sequential steps: patient screening, apheresis, bridging therapy (as needed), CAR-T infusions and follow up for up to two years. If the safety and tolerability are acceptable and recommended phase 2 dose (RP2D) is determined from the dose escalation stage, dose expansion will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects have been fully informed of the possible risks and benefits of participating in this study and have voluntarily signed the informed consent form (ICF).
2. Age: 18-70 years (including 18 and 70 years).
3. ECOG 0-1.
4. With an expected survival of more than 3 months.
5. Patients with histologically or cytologically confirmed locally advanced or metastatic "BT-001 positive" solid tumors. IHC should be within 6 months of apheresis, but maybe extended.
6. Preference for patients who have failed first- or second-line therapy.
7. Having measurable lesions according to RECIST 1.1 (or the latest version).
8. Maximum tumor size less than 4 cm according to RECIST 1.1 (or the latest version).
9. Having sufficient bone marrow, liver, kidney, and lung functions (based on the normal value of the clinical trial sites).

   * ANC and PLT ≥ LLN.
   * Without liver metastases, ALT, AST, or ALP ≤ 2.5×upper limit of normal (ULN); with liver metastases, ALT, AST, or ALP ≤ 5×ULN.
   * Serum creatinine (ScR) ≤ 1.5×ULN, or creatinine clearance > 50 mL/min (calculated according to Cockcroft Gault formula).
   * International normalized ratio (INR) ≤ 1.5×ULN, APTT ≤ 1.5×ULN.
   * Adequate oxygen saturation (≥ 95%) can be maintained without oxygen inhalation.
10. Male or female patients of childbearing potential agree to use effective methods of contraception (such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, and intrauterine devices) during the study period and within 1 year after infusion.

Exclusion Criteria:

1. Patients who have received the following anti-tumor treatments prior to apheresis:

   1. Cytotoxic therapy within 14 days or 28 days (for chemotherapy with high lymphocytic toxicity such as bendamustine, cyclophosphamide, ifosfamide, fludarabine, cladribine, etc.).
   2. Small molecule targeted therapy within 14 days or at least 5 half-lives, whichever is longer.
   3. Therapy with monoclonal antibody within 21 days including cetuximab.
   4. Therapy with immune checkpoint inhibitors and/or Avastin within 30 days of apheresis.
   5. Immunomodulatory therapy within 14 days.
   6. Radiotherapy within 14 days of apheresis.
   7. Traditional Chinese medicine with anti-tumor indications within 14 days of apheresis.
   8. Investigational agents or treatment within 28 days of apheresis.
   9. Previously treated with CAR-T/TCR-T cells and/or vaccine within 28 days of apheresis.
2. Previously treated with any BT-001-targeted therapy.
3. Brain metastases with central nervous system symptoms.
4. Pregnant (positive pregnancy test prior to dosing) or breast-feeding.
5. Allergic or suspected allergic reaction to any drug and related excipients specified in protocol, e.g., camelid antibody, pre-infusion medication (acetaminophen and diphenhydramine), serum albumin, tocilizumab (or biosimilars of tocilizumab that have been approved for CRS indication), Erbitux/ cetuximab, dimethyl sulfoxide (DMSO), and dextran 40.
6. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B virus (HBV) deoxyribonucleic acid (DNA) > 100IU/mL or lower limit of the research center [Only when the detection limit of the research center is higher than 100IU/mL]), or patients with positive HCV antibody.
7. Patients with a history of immunodeficiency, including those who are HIV-positive, or patients with other acquired or congenital immune deficiency, or a history of organ transplantation.
8. Patients with concomitant or previous history of interstitial lung disease or interstitial pneumonia; presence of multiple metastatic lesions in the lungs or a single metastatic lesion ≥ 3 cm in length; patients with inflammation in the lungs or have received extensive radiotherapy.
9. Patients with uncontrolled active infection based on the investigator's judgment.
10. Patients who underwent major surgery within 2 weeks prior to apheresis and not fully recovered.
11. The toxicity of previous anti-cancer therapy, including immunotherapy has not returned to less than or equal to Grade 1 as specified in CTCAE v5.0 or the latest version (except for hair loss, Grade 2 peripheral neuropathy, and stable hypothyroidism treated with hormone replacement therapy).
12. Patients with a history of acute myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack within 6 months prior to the enrollment, or with NYHA Class 2 or higher congestive heart failure.
13. Patients with chronic diseases requiring treatment with systemic corticosteroids or other immunosuppressants, received systemic corticosteroids (≥ 70 mg prednisone or equivalent dose of other corticosteroids) or other immunosuppressants within 7 days before apheresis, except for the following cases: local, ocular, intra-articular, intranasal, and inhaled glucocorticoid treatment; short term use of glucocorticoids for preventive treatment (such as prevention of contrast medium allergy).
14. Patients with autoimmune diseases.
15. Patients with Crohn's Disease.
16. Patients with a history of uncontrollable mental illness.
17. Any condition in which the investigator considers that the subject is not suitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of B4T2-001 CAR-T will be assessed by the incidence of serious adverse events (SAEs), incidence and severity of adverse events (AEs). | 2 years after B4T2-001 CAR-T
  Multiple infusions of B4T2-001 CAR-T.
To determine the MTD and RP2D of B4T2-001 CAR-T | 2 years after B4T2-001 CAR-T
  The MTD will be determined based on the occurrence of the DLTs according to dose escalation design. RP2D will be defined based on MTD, safety, PK, and preliminary efficacy data.

SECONDARY OUTCOMES:
PK parameters: maximum concentration (Cmax) | Blood sampling for PK will be performed till 2 years after B4T2-001 CAR-T
  Maximum concentration (Cmax) with the immunoanalytical method.
PK parameters: time of peak concentration (Tmax) | Blood sampling for PK will be performed till 2 years after B4T2-001 CAR-T
  Time to peak concentration (Tmax) with the immunoanalytical method.
PK parameters: the last measurable time point (Tlast) | Blood sampling for PK will be performed till 2 years after B4T2-001 CAR-T
  The last measurable time point (Tlast) with the immunoanalytical method.
PK parameters: area under the curve (AUCs) | Blood sampling for PK will be performed till 2 years after B4T2-001 CAR-T
  Area under the curve (AUCs)with the immunoanalytical method.
Overall response rate (ORR) after administration | 2 years after B4T2-001 CAR-T
  ORR is defined as the proportion of subjects who achieve CR or PR after treatment via B4T2-001 CAR T, and the objective tumor response rate will be calculated for patients with measurable disease per by RECIST 1.1 (or the latest version) supplemented by iRecist.
Duration of Response (DOR) after administration | 2 years after B4T2-001 CAR-T
  DOR is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (by RECIST 1.1 (or the latest version) supplemented by iRecist) of the responders (who achieve PR or better response).
Progress Free Survival (PFS) after administration | 2 years after B4T2-001 CAR-T
  PFS is defined as the time from the date of first infusion of the B4T2-001 to the first documented disease progression (according to by RECIST 1.1 (or the latest version) supplemented by iRecist) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | 2 years after B4T2-001 CAR-T
  OS is defined as the time from the date of first infusion of B4T2-001 CAR-T to death of the subject.

OTHER OUTCOMES:
Blood cytokine levels include interleukin 6 (IL-6), IL-2, IL-4, IL-8, IL-10, TNF-α, and INF-γ with ELISA or equivalent method | Blood sampling for cytokine measurement will be performed at planned time points till 2 years after B4T2-001 CAR-T.
  Concentration and kinetics of multiple blood cytokines including (IL-6), IL-2, IL-4, IL-8, IL-10, TNF-α, and INF-γ which have the same unit of measure, and using ELISA or equivalent before and after CAR-T and will be evaluated according to actual blood sampling time points.
H score (0-300) | Planned time points till 2 years after B4T2-001 CAR-T
  Explore and evaluate histology before and possibly after CAR-T for expression of BT-001 antigen on the tumor by immunohistochemistry (IHC) to determine the score intensity. "BT-001 positive" refers to a staining of H score of > 150 and preference will be patients with H score of > 200. H score (0-300) will be calculated. High scores are desired.
Overall IHC Score (0-4) | Planned time points till 2 years after B4T2-001 CAR-T
  Explore and evaluate histology before and possibly after CAR-T for expression of BT-001 antigen on the tumor by IHC to evaluate the score intensity. "BT-001 positive" refers to an IHC score ≥ 3 and preference will be patients with an IHC score of 4. Overall IHC Score (0-4) will be calculated. High scores are desired.
The percentage of BT-001 positive stained tumor | Planned time points till 2 years after B4T2-001 CAR-T
  Explore and evaluate histology before and possibly after CAR-T for heterogeneity of expression of BT-001 antigen on the tumor.
Exploratory tumor biomarker evaluation | Planned time points till 2 years after B4T2-001 CAR-T
  Explore and evaluate tumor markers, such as CEA before and possibly after CAR-T.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, PhD, Principal Investigator — Shanghai East Hospital
Locations (2):
- China (2):
  - Shanghai East Hospital, Shanghai, China/Shanghai
  - Shanghai Artemed Hospital, Shanghai, China/Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Kershaw MH, Westwood JA, Darcy PK. Gene-engineered T cells for cancer therapy. Nat Rev Cancer. 2013 Aug;13(8):525-41. doi: 10.1038/nrc3565. PMID 23880905
- [Background] Kochenderfer, J.N., et al., Effective Treatment Of Chemotherapy-Refractory Diffuse Large B-Cell Lymphoma With Autologous T Cells Genetically-Engineered To Express An Anti-CD19 Chimeric Antigen Receptor. Blood, 2013. 122(21): p. 168-168.
- [Background] Thompson JA, Schneider BJ, Brahmer J, Achufusi A, Armand P, Berkenstock MK, Bhatia S, Budde LE, Chokshi S, Davies M, Elshoury A, Gesthalter Y, Hegde A, Jain M, Kaffenberger BH, Lechner MG, Li T, Marr A, McGettigan S, McPherson J, Medina T, Mohindra NA, Olszanski AJ, Oluwole O, Patel SP, Patil P, Reddy S, Ryder M, Santomasso B, Shofer S, Sosman JA, Wang Y, Zaha VG, Lyons M, Dwyer M, Hang L. Management of Immunotherapy-Related Toxicities, Version 1.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Apr;20(4):387-405. doi: 10.6004/jnccn.2022.0020. PMID 35390769
- [Background] Jo Y, Ali LA, Shim JA, Lee BH, Hong C. Innovative CAR-T Cell Therapy for Solid Tumor; Current Duel between CAR-T Spear and Tumor Shield. Cancers (Basel). 2020 Jul 28;12(8):2087. doi: 10.3390/cancers12082087. PMID 32731404
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Del Bufalo F, De Angelis B, Caruana I, Del Baldo G, De Ioris MA, Serra A, Mastronuzzi A, Cefalo MG, Pagliara D, Amicucci M, Li Pira G, Leone G, Bertaina V, Sinibaldi M, Di Cecca S, Guercio M, Abbaszadeh Z, Iaffaldano L, Gunetti M, Iacovelli S, Bugianesi R, Macchia S, Algeri M, Merli P, Galaverna F, Abbas R, Garganese MC, Villani MF, Colafati GS, Bonetti F, Rabusin M, Perruccio K, Folsi V, Quintarelli C, Locatelli F; Precision Medicine Team-IRCCS Ospedale Pediatrico Bambino Gesu. GD2-CART01 for Relapsed or Refractory High-Risk Neuroblastoma. N Engl J Med. 2023 Apr 6;388(14):1284-1295. doi: 10.1056/NEJMoa2210859. PMID 37018492
- [Background] Qi C, Gong J, Li J, Liu D, Qin Y, Ge S, Zhang M, Peng Z, Zhou J, Cao Y, Zhang X, Lu Z, Lu M, Yuan J, Wang Z, Wang Y, Peng X, Gao H, Liu Z, Wang H, Yuan D, Xiao J, Ma H, Wang W, Li Z, Shen L. Claudin18.2-specific CAR T cells in gastrointestinal cancers: phase 1 trial interim results. Nat Med. 2022 Jun;28(6):1189-1198. doi: 10.1038/s41591-022-01800-8. Epub 2022 May 9. PMID 35534566
- [Background] Gauthier J, Bezerra ED, Hirayama AV, Fiorenza S, Sheih A, Chou CK, Kimble EL, Pender BS, Hawkins RM, Vakil A, Phi TD, Steinmetz RN, Jamieson AW, Bar M, Cassaday RD, Chapuis AG, Cowan AJ, Green DJ, Kiem HP, Milano F, Shadman M, Till BG, Riddell SR, Maloney DG, Turtle CJ. Factors associated with outcomes after a second CD19-targeted CAR T-cell infusion for refractory B-cell malignancies. Blood. 2021 Jan 21;137(3):323-335. doi: 10.1182/blood.2020006770. PMID 32967009
- [Background] Hines MR, Knight TE, McNerney KO, Leick MB, Jain T, Ahmed S, Frigault MJ, Hill JA, Jain MD, Johnson WT, Lin Y, Mahadeo KM, Maron GM, Marsh RA, Neelapu SS, Nikiforow S, Ombrello AK, Shah NN, Talleur AC, Turicek D, Vatsayan A, Wong SW, Maus MV, Komanduri KV, Berliner N, Henter JI, Perales MA, Frey NV, Teachey DT, Frank MJ, Shah NN. Immune Effector Cell-Associated Hemophagocytic Lymphohistiocytosis-Like Syndrome. Transplant Cell Ther. 2023 Jul;29(7):438.e1-438.e16. doi: 10.1016/j.jtct.2023.03.006. Epub 2023 Mar 9. PMID 36906275
- [Background] Jain MD, Smith M, Shah NN. How I treat refractory CRS and ICANS after CAR T-cell therapy. Blood. 2023 May 18;141(20):2430-2442. doi: 10.1182/blood.2022017414. PMID 36989488
- [Background] Alvi RM, Frigault MJ, Fradley MG, Jain MD, Mahmood SS, Awadalla M, Lee DH, Zlotoff DA, Zhang L, Drobni ZD, Hassan MZO, Bassily E, Rhea I, Ismail-Khan R, Mulligan CP, Banerji D, Lazaryan A, Shah BD, Rokicki A, Raje N, Chavez JC, Abramson J, Locke FL, Neilan TG. Cardiovascular Events Among Adults Treated With Chimeric Antigen Receptor T-Cells (CAR-T). J Am Coll Cardiol. 2019 Dec 24;74(25):3099-3108. doi: 10.1016/j.jacc.2019.10.038. PMID 31856966
- [Background] Ghosh AK, Chen DH, Guha A, Mackenzie S, Walker JM, Roddie C. CAR T Cell Therapy-Related Cardiovascular Outcomes and Management: Systemic Disease or Direct Cardiotoxicity? JACC CardioOncol. 2020 Mar 17;2(1):97-109. doi: 10.1016/j.jaccao.2020.02.011. eCollection 2020 Mar. PMID 34396213
- [Background] Haerizadeh F, Jiang H, Cooper L. Selective recognition of over-expressed self-antigens in solid tumors using calibrated CAR-T therapy. Journal of Clinical Oncology 2023 41:16_suppl, 2540-2540